CLINICAL TRIAL: NCT00932295
Title: Evaluating the Acute Effects of Electronic Nicotine Delivery Devices Marketed to Smokers.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HM11820; R01CA103827 (NIH); R01CA120142 (NIH)
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Smoking
Keywords: tobacco; cigarette; nicotine
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Own brand cigarette (Active Comparator): 10 puffs from the participants own brand brand of cigarette (lit; 30 second inter puff interval)
  Interventions: Other: OB
- Sham smoking (Sham Comparator): 10 puffs from the participants own brand brand of cigarette (NOT lit; 30 second inter puff interval)
  Interventions: Other: Sham smoking
- Electronic cigarette Version One C7 (Experimental): 10 puffs from a so-called "electronic cigarette" named CROWN SEVEN (16 mg cartridge; 30 second inter puff interval)
  Interventions: Other: CROWN SEVEN
- Electronic cigarette version 2: NJ (Experimental): 10 puffs from a so-called "electronic cigarette" named NJOY (16 mg cartridge; 30 second inter puff interval)
  Interventions: Other: NJOY

INTERVENTIONS:
Other: OB — 10 puffs from the participants own brand brand of cigarette (lit; 30 second inter puff interval)
  Arms: Own brand cigarette
Other: Sham smoking — 10 puffs from the participants own brand brand of cigarette (NOT lit; 30 second inter puff interval)
  Arms: Sham smoking
Other: CROWN SEVEN — 10 puffs from a so-called "electronic cigarette" named CROWN SEVEN (16 mg cartridge; 30 second inter puff interval)
  Arms: Electronic cigarette Version One C7
Other: NJOY — 10 puffs from a so-called "electronic cigarette" named NJOY(16 mg cartridge; 30 second inter puff interval)
  Arms: Electronic cigarette version 2: NJ

SUMMARY:
The study's aim is to develop a clinical model that can be used to measure the nicotine delivery and tobacco/nicotine abstinence-suppressing capability of electronic devices that are marketed as a means to deliver nicotine to cigarette smokers. The study will compare the nicotine delivery, cardiovascular effects, and tobacco withdrawal suppressing effects of two devices currently marketed in the U.S.: Crown Seven and NJOY. Specifically, the effects of these devices will be compared with the effects of own brand cigarettes (positive control), and an abstinence condition (sham smoking; puffing from an unlit cigarette). The primary hypothesis is that the nicotine delivery, withdrawal suppression, and other effects of electronic devices marketed as a means to deliver nicotine to smokers can be measured during a period of acute exposure.

DETAILED DESCRIPTION:
Potential reduced exposure products (PREPs) are being developed and marketed by the tobacco industry in an attempt to reduce some of the risks involved in tobacco use (see Breland et al., 2002b). Evaluating the effects of these products is crucial to public health, as past industry-sponsored efforts at harm reduction (e.g., so-called "light" and "ultra-light" cigarettes) were not evaluated and failed to reduce carbon monoxide (CO), nicotine, and carcinogen exposure in smokers; these efforts thus failed to reduce the harms of smoking (Stratton et al., 2001). This study is part of an on-going, NIH-funded program of research to develop a science-based model that uses outcome measures relevant to evaluating current tobacco industry-sponsored smoking harm reduction efforts systematically and efficiently.

ELIGIBILITY:
Inclusion Criteria:

Participants must be healthy, between 18 and 55 years of age, and report a cigarette intake of > 15 cig/day for at least 1 year. They must provide an afternoon screening CO level of > 15 ppm at intake. They must also provide a urine sample for cotinine analysis, and receive a result of at least 4 on the urine immunoassay test strip scale (possible range = 0-6) at intake.

Exclusion Criteria:

Exclusion criteria include: history of chronic health problems or psychiatric conditions, breastfeeding, or pregnancy (assessed by urinalysis). Individuals who report current attempts to quit smoking, previous experience with Crown Seven or NJOY. Individuals who report alcohol or marijuana use greater than 20 days within the last 30 days, or recent illicit drug use such as cocaine or heroin. Women reporting active menopause will be excluded (menopause may cause tobacco/nicotine withdrawal-like symptoms, such as depression, Parry et al., 2001).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Plasma nicotine concentration (ng/ml) | baseline, 5, 15, 30, and 45 minutes post-use

SECONDARY OUTCOMES:
Heart rate | continuous
Withdrawal suppression (subjective measure) | baseline and 5, 15, 30, and 45 minutes post-use

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eissenberg, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Clinical Behavioral Pharmacology Laboratory, Richmond, Virginia, United States

REFERENCES:
- [Background] Cobb CO, Weaver MF, Eissenberg T. Evaluating the acute effects of oral, non-combustible potential reduced exposure products marketed to smokers. Tob Control. 2010 Oct;19(5):367-73. doi: 10.1136/tc.2008.028993. Epub 2009 Apr 2. PMID 19346218
- [Background] Gray JN, Breland AB, Weaver M, Eissenberg T. Potential reduced exposure products (PREPs) for smokeless tobacco users: clinical evaluation methodology. Nicotine Tob Res. 2008 Sep;10(9):1441-8. doi: 10.1080/14622200802323258. PMID 19023835
- [Background] Blank MD, Sams C, Weaver MF, Eissenberg T. Nicotine delivery, cardiovascular profile, and subjective effects of an oral tobacco product for smokers. Nicotine Tob Res. 2008 Mar;10(3):417-21. doi: 10.1080/14622200801901880. PMID 18324559
- [Background] Breland AB, Kleykamp BA, Eissenberg T. Clinical laboratory evaluation of potential reduced exposure products for smokers. Nicotine Tob Res. 2006 Dec;8(6):727-38. doi: 10.1080/14622200600789585. PMID 17132520
- [Background] Breland AB, Evans SE, Buchhalter AR, Eissenberg T. Acute effects of Advance: a potential reduced exposure product for smokers. Tob Control. 2002 Dec;11(4):376-8. doi: 10.1136/tc.11.4.376. PMID 12432165